CLINICAL TRIAL: NCT07271550
Title: Cross-cultural Adaptation and Validation of the Nottingham Assessment of Functional Footcare (NAFF) Questionnaire Among Arabic-speaking Adults With Diabetes in Tunisia
Brief Title: NAFF Arabic Validation Study
Status: Completed | Type: Observational
Sponsor: Faculty of Medicine, Sousse (Other)
Responsible Party: Principal Investigator, Emna Taghouti, Doctorante, Investigateur Principal, Faculty of Medicine, Sousse
Other Study IDs: NAFF-A
Record Dates: First submitted 2025-08-29; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Diabetic Foot Disease; Behavior; Self Care; Questionnaire and Survey
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate a new Arabic version of the NAFF questionnaire, which measures foot care behaviors in adults with type 2 diabetes. Participants are adults with type 2 diabetes who will complete the questionnaire online. The study will assess how reliable and valid the Arabic version is, helping healthcare providers identify risky foot care behaviors and improve patient education.

DETAILED DESCRIPTION:
This study is a cross-sectional validation of the NAFF questionnaire translated into Arabic. Adult patients with type 2 diabetes will be recruited from endocrinology outpatient clinic in Sousse. Participants will complete the Arabic NAFF online. Primary outcomes include assessment of reliability (internal consistency, test-retest) and validity (construct and criterion validity). Secondary outcomes include the relationship between foot care behaviors and demographic or clinical factors. All participants will provide informed consent electronically. The study protocol was approved by the Ethics Committee of the Faculty of Medicine, Sousse. Data will be analyzed using descriptive and inferential statistics to evaluate the psychometric properties of the Arabic NAFF..

ELIGIBILITY:
Inclusion Criteria:

* Adults diagnosed with type 2 diabetes mellitus
* Age 26-65 years
* Ability to read and understand Arabic
* Receiving regular follow-up care at the endocrinology outpatient clinic

Exclusion Criteria:

* Cognitive impairments affecting comprehension or self-care activities
* Physical disabilities hindering self-care activities
* Presence of active foot ulcers at time of enrollment
* Bilateral lower-limb amputations

Ages: 26 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Translation and adaptation | 01/06/ 2021-31/07/ 2021 (2 months)
  Translation, cultural adaptation, and assessment of content validity through expert panel evaluation using a 4-point relevance scale. Content validity index calculated by dividing items rated 3-4 by total items (n=29). Values ≥0.80 considered acceptable.
Descriptive data | 01/08/2021 to 28/11/2021 (4 months)
  Participants were asked to complete the NAFF-A questionnaire in the waiting room before clinical consultation. Demographic and clinical data were collected from medical records in collaboration with attending physicians, including gender, age, educational level, residence, diabetes duration, HbA1c levels, and history of ulceration or amputation.
Test-Retest Reliability of NAFF-A (Intraclass Correlation Coefficient) | Test-retest interval of 10-14 days between initial assessment and follow-up assessment.
  Assessment of temporal stability of the NAFF-A using intraclass correlation coefficient (ICC) between test and retest administrations. Values ≥0.70 indicate good reliability, with higher values indicating better temporal stability.

SECONDARY OUTCOMES:
Internal consistency | At the end of data collection
  Assessment of internal consistency reliability of the Arabic version of the Nottingham Assessment of Functional Footcare questionnaire using Cronbach's alpha coefficient. Acceptable range is 0.70-0.95, with higher values indicating better internal consistency.
Criterion Validity - Correlation with Educational Level | At the end of data collection
  Spearman's correlation coefficient between NAFF-A total scores and participant educational level (primary, secondary, university). Positive correlation expected based on literature showing higher education associated with better self-care behaviors.
Criterion Validity - Correlation with HbA1c Levels | At the end of data collection
  Spearman's correlation coefficient between NAFF-A total scores and glycated hemoglobin (HbA1c) levels. Negative correlation expected as better foot care behaviors should be associated with better glycemic control.
Criterion Validity - Correlation with Ulceration Risk Stratification | At the end of data collection
  Spearman's correlation coefficient between NAFF-A total scores and ulceration risk grades (0-3 scale based on IWGDF guidelines). Negative correlation expected as better foot care behaviors should be associated with lower ulceration risk.

CONTACTS AND LOCATIONS:
Locations (1):
- Farhat Hached University Hospital, Endocrinology Department, Sousse, Sousse Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared publicly due to ethical constraints and participant privacy protections as per the Ethics Committee approval (CEFMS 81/2021) and Tunisian data protection regulations. Aggregate data and statistical results are available through the published manuscript. Researchers interested in collaboration may contact the principal investigator to discuss potential data sharing arrangements that comply with ethical and regulatory requirements.